CLINICAL TRIAL: NCT03675776
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of Rapastinel as Monotherapy in Patients With Major Depressive Disorder
Brief Title: Study of Rapastinel as Monotherapy in Patients With Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to stop the program.
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAP-MD-30; 2018-000060-29 (EudraCT Number)
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Depressive Disorder, Major
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rapastinel 450mg (Experimental): Rapastinel (prefilled syringe, weekly intravenous IV administration).
  Interventions: Drug: Rapastinel
- Rapastinel 225mg (Experimental): Rapastinel (prefilled syringe, weekly intravenous IV administration).
  Interventions: Drug: Rapastinel
- Placebo (Placebo Comparator): Placebo (prefilled syringe, weekly IV administration).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapastinel — Rapastinel (prefilled syringe, weekly intravenous IV administration).
  Arms: Rapastinel 225mg; Rapastinel 450mg
Drug: Placebo — Placebo (prefilled syringe, weekly IV administration).
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy, safety, and tolerability of 225 milligrams (mg) and 450 milligrams (mg) of Rapastinel, compared to placebo in participants with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD
* Current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Visit 1
* Treatment naive in the current episode or have inadequate response to 1-3 antidepressant therapies given at adequate dose and duration in the current episode
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test

Exclusion Criteria:

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1
* Lifetime history of meeting DSM-5 criteria for:

  1. Schizophrenia spectrum or other psychotic disorder
  2. Bipolar or related disorder
  3. Major neurocognitive disorder
  4. Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
  5. Dissociative disorder
  6. Posttraumatic stress disorder
  7. MDD with psychotic features
* Significant suicide risk, as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (23):
- Bugát Pál Hospital, Clinexpert, Gyöngyös, Hungary
- Japan (15):
  - Himorogi Psychiatric Institute, Ichigayatamachi
  - Kishiro Mental Clinic, Kawasaki-shi
  - Tatsuta Clinic, Kobe
  - Medical corporation Sato-Kai Yuge Hospital, Kumamoto
  - Sagaarashiyama-Tanaka Clinic, Kyoto
  - Senzoku psychosomatic Medicine Clinic, Meguro-ku
  - Higashi Sapporo Mental Clinic, Sapporo
  - Sangenjaya Neurology- Psychosomatic Clinic, Setagaya-ku
  - Yoyogi Mental Clinic, Shibuya-ku
  - Maynds Tower Mental Clinic, Shibuya-ku
  - Himeno Tomomi Clinic, Shinagawa-ku
  - Shinjuku Research Park Clinic, Shinjuku-ku
  - Ohwa Mental Clinic, Toshima-ku
  - Okehazama Hospital Fujita Kokoro Care Center, Toyoake
  - Yokohama Onoecho Clinic, Yokohama
- Centrum Medyczne Luxmed Sp.z o.o., Lublin, Poland
- Russia (2):
  - Federal State Budgetary Research Institution "Mental Health Science Center", Moscow
  - Yaroslavl Regional Psychiatric Hospital, Yaroslavl
- Slovakia (4):
  - MENTUM, s.r.o., Bratislava
  - Vavrusova Consulting s.r.o. Neštátna Psychiatrická ambulancia, Bratislava
  - Liptovská nemocnica s poliklinikou MUDr. Ivana Stodolu Liptovský Mikuláš, Liptovský Mikuláš
  - Psycholine s.r.o., Rimavská Sobota

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://www.allerganclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 68 participants were screened for eligibility; 50 participants randomized to receive double-blind treatment.
Period: Double Blind Treatment Period
Arm/Group | Placebo | Rapastinel 225mg | Rapastinel 450mg
Started | 15 | 17 | 18
Completed | 9 | 11 | 10
Not Completed | 6 | 6 | 8
Not completed — Study Terminated by Sponsor | 5 | 6 | 8
Not completed — Lack of Efficacy | 1 | 0 | 0
Period: Safety Follow-up Period
Arm/Group | Placebo | Rapastinel 225mg | Rapastinel 450mg
Started | 6 | 8 | 7
Completed | 6 | 8 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat (mITT) Population consisted of all patients in the Safety Population who had at least 1 postbaseline assessment of the MADRS total score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rapastinel 225mg | Rapastinel 450mg | Total
Number analyzed (Participants) | 15 | 17 | 18 | 50
Age, Continuous [Median (Standard Deviation); unit: Years] | 42.4 (10.36) | 44.7 (10.83) | 43.2 (11.06) | 43.5 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 7 | 27
  Male | 8 | 4 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 17 | 18 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 7 | 9 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 10 | 9 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 73.86 (13.14) | 69.58 (16.52) | 70.32 (15.72) | 71.13 (15.09)
Height [Mean (Standard Deviation); unit: cm] | 169.27 (10.68) | 163.77 (5.90) | 168.04 (6.36) | 166.96 (7.97)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.83 (4.41) | 25.85 (5.50) | 24.82 (5.09) | 25.47 (4.97)
Montgomery-Asberg Depression Rating Scale (MADRS) total score at baseline [Mean (Standard Deviation); unit: Score on a scale] — The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement
  Score on a scale | 34.5 (4.34) | 35.2 (4.78) | 34.8 (4.72) | 34.9 (4.54)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at End of Double-blind Treatment (End of Week 6).
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
Time Frame: Baseline to end of Week 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rapastinel 225mg | Rapastinel 450mg
Number analyzed (Participants) | 15 | 17 | 18
Score on a scale | -11.3 (9.06) | -21.3 (10.31) | -12.9 (11.36)

2. Secondary Outcome: Change From Baseline in MADRS Total Score at 1 Day After First Dose of Treatment
Description: as for outcome 1
Time Frame: Baseline to 1 Day post-first dose
Population: The Modified Intent-to-Treat (mITT) Population consists of all patients in the Safety Population who had at least 1 postbaseline assessment of the MADRS total score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Rapastinel 225mg | Rapastinel 450mg
Number analyzed (Participants) | 15 | 17 | 18
Score on a scale | -6.7 (5.36) | -7.4 (9.10) | -6.4 (9.11)

ADVERSE EVENTS:
Time Frame: The study consisted of a 6 week double-blind treatment period, followed by a 2-week safety follow-up period.
Description: Safety Population consists of all randomized patients who received at least 1 dose of randomized investigational product (IP).
Arm/Group | Placebo | Rapastinel 225mg | Rapastinel 450mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 6/15 | 1/17 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Rapastinel 225mg (N=17) | Rapastinel 450mg (N=18)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to study termination, the target number of participants needed to achieve target power and statistically reliable results was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT03675776/SAP_000.pdf
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03675776/Prot_001.pdf